CLINICAL TRIAL: NCT03803891
Title: Multicenter Prospective Study of Endoscopic Full-thickness Resection (EFTR) in Colon Using Over-the-scope-clip (OTSC)
Brief Title: Endoscopic Full-Thickness Resection In Colon
Acronym: EFTRICOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other); Hospital de Sant Joan Despí Moisès Broggi (Other); Complejo Hospitalario de Navarra (Other); Hospital Clínico Universitario de Santiago de Compostela (Unknown); Hospital Provincial de Castellon (Other); Althaia Xarxa Assistencial Universitària de Manresa (Other); Hospital Mutua de Terrassa (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital San Carlos, Madrid (Other); Hospital Universitario 12 de Octubre (Other); Hospital General de Ciudad Real (Other); Hospital General Universitario Elche (Other); Hospital Universitario Central de Asturias (Other); Hospital Clinic of Barcelona (Other); Quironsalud (Other); Hospital Universitario La Paz (Other); Centro Medico Teknon (Other); Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, HugoUchima, Medical Specialist (gastroenterologist, MD), Fundació Institut Germans Trias i Pujol
Other Study IDs: HU-EMPRET
Record Dates: First submitted 2018-12-17; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Colon Neoplasm, Malignant; Colo-rectal Cancer; Colonic Cancer; Colonic Adenoma; Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenocarcinoma; Colon Polyp; Colon Lesion; Colon Neoplasm
Keywords: Endoscopic resection; Colonoscopy; Full-thickness resection
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic full-thickness resection: Patients with neoplastic lesions less than 30mm unresectable en bloc by other less invasive endoscopic techniques, including lesions suggestive of T1 colorectal cancer, subepithelial tumors, lesions with diverticular involvement, lesions with no-lifting sign (recurrent, incomplete prior resection or untreated lesions).
  Interventions: Procedure: Endoscopic full-thickness resection

INTERVENTIONS:
Procedure: Endoscopic full-thickness resection — Endoscopic full-thickness resection (EFTR) with Over-The-Scope-Clip in colorectal lesions

SUMMARY:
Endoscopic full-thickness resection (EFTR) in the colon using an over-the-scope clip (OTSC) as a closure mechanism is a recent technique that allows the endoscopic resection of colonic lesions that are poor candidates for conventional endoscopic resection techniques. The aim is to study the safety and efficacy of EFTR in colon.

DETAILED DESCRIPTION:
Early detection and endoscopic resection of early neoplastic lesions in colon can prevent the development of colon cancer.

The classic endoscopic mucosal resection technique and the submucosal dissection technique require the creation of a submucosal "cushion" by injecting crystalloid substances or colloids. However, these advanced techniques have technical limitations when facing a lesion that presents poor lifting or non-lifting at all as it might be observed in scarring or fibrotic lesions

Endoscopic full-thickness resection (EFTR) in the colon using an over-the-scope clip (OTSC) is a recent technique that does not require the injection of a submucosal solution and allows a resection of colonic lesions of up to approximately 30 mm, en bloc, allowing a correct histological study of the sample, to confirm its complete resection with adequate deep margins, evaluation of the level of invasion and lymphovascular involvement.

EFTR with OTSC allows a colonic wall full-thickness resection, by the deployment of an over-the-scope clip before the resection of the lesion to prevent perforation. The steps of the technique are: face the lesion and marking the borders, insertion of the scope with the kit (consisting of a cap with an integrated snare and OTSC), grasping and pulling the lesion into the cap, deploy the over-the-scope-clip (OTSC) and closing the integrated snare and resect.

This is a multicenter observational study on the efficacy and safety of EFTR with OTSC in colon.

The clinical, endoscopic and histological data are collected prospectively in all cases of EFTR performed in the participant centers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) of both sexes.
* Colonic lesions less than 30mm unresectable en-bloc by other less invasive endoscopic techniques, including lesions suggestive of T1, subepithelial tumors, lesions with diverticular involvement, lesions with no-lifting signs (recurrent, incomplete prior resection or untreated).
* Patients who give their written informed consent for the procedure and for the study.

Exclusion Criteria:

* Refusal to grant informed consent.
* Neoplastic lesions of the colon with evidence of advanced stage (for example, lymph node involvement) or more than 3 cm in greatest diameter.
* Any medical, psychological, geographical, or social problem that is significant and uncontrolled that may interfere with the patient's participation in the study or that does not allow adequate follow-up and adherence to the protocol and evaluation of the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo a endoscopic full-thickness resection for colonic lesions who meet the inclusion criteria will be included consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Through study completion, an average of 1 year
  Percentage of complete en-bloc resection of the lesion without macroscopic residual tissue after completing the endoscopic full-thickness resection

SECONDARY OUTCOMES:
Major adverse events | 3 months
  Percentage of procedure-associated major adverse events: bleeding and/or perforation
Histologically confirmed full-thickness resection | 30 days
  Histologically confirmed full-thickness resection

CONTACTS AND LOCATIONS:
Overall Officials: Hugo I. Uchima Koecklin, MD, Principal Investigator — Medical researcher
Locations (15):
- Spain (15):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Fundació Althaia, Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Quirónsalud Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt A, Meier B, Caca K. Endoscopic full-thickness resection: Current status. World J Gastroenterol. 2015 Aug 21;21(31):9273-85. doi: 10.3748/wjg.v21.i31.9273. PMID 26309354
- [Background] Uchima H, Barquero D, Fernandez A, Mata A, Huertas C, Figa M, Hombrados M, Espinos JC. Su1638 Early Discharge After Endoscopic Full-Thickness Resection in the Colorectum. Gastrointest Endosc. 2017;85:5, AB375
- [Background] Schmidt A, Beyna T, Schumacher B, Meining A, Richter-Schrag HJ, Messmann H, Neuhaus H, Albers D, Birk M, Thimme R, Probst A, Faehndrich M, Frieling T, Goetz M, Riecken B, Caca K. Colonoscopic full-thickness resection using an over-the-scope device: a prospective multicentre study in various indications. Gut. 2018 Jul;67(7):1280-1289. doi: 10.1136/gutjnl-2016-313677. Epub 2017 Aug 10. PMID 28798042
- [Background] Backes Y, Kappelle WFW, Berk L, Koch AD, Groen JN, de Vos Tot Nederveen Cappel WH, Schwartz MP, Kerkhof M, Siersema PD, Schroder R, Tan TG, Lacle MM, Vleggaar FP, Moons LMG; T1 CRC Working Group. Colorectal endoscopic full-thickness resection using a novel, flat-base over-the-scope clip: a prospective study. Endoscopy. 2017 Nov;49(11):1092-1097. doi: 10.1055/s-0043-114730. Epub 2017 Jul 28. PMID 28753696